CLINICAL TRIAL: NCT05166291
Title: The Effect of Needle-free Injection System Versus Traditional Anesthesia on Pain Perception During Palatal Infiltration Anesthesia in Children: a Randomized Clinical Trial
Brief Title: The Effect of Needle-free Injection System During Palatal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Kaya, Principal Investigator, Okan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E.617498811-000-1065232
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Pediatric Anesthesia; Local Anesthesia
Keywords: needle-free injection system; pain perception

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional anesthesia (TA) (Experimental): traditional anesthesia
  Interventions: Other: traditional anesthesia
- comfort-in injection system (CIS) (Experimental): comfort-in injection system (CIS)
  Interventions: Device: Comfort-in injection system

INTERVENTIONS:
Device: Comfort-in injection system — local anesthesia applyed with comfort-in injection system
  Other Names: dental syringe
  Arms: comfort-in injection system (CIS)
Other: traditional anesthesia — local anesthesia applyed with dental syringe
  Arms: traditional anesthesia (TA)

SUMMARY:
Needle-free injection systems can contribute to the prevention of needle-related pain during palatal infiltration anesthesia (PIA) in children. Research with this topic on children is required.The purpose of this clinical study was to evaluate the effectiveness of the needle-free system versus traditional anesthesia on pain perception during PIA in children.The study was designed as a randomized, controlled cross-over clinical study with 48 children aged 6 to 12 years requiring dental treatment with PIA in bilateral maxillary primary molars. It has been revealed that the application of a needle-free system during PIA ensured a decrease in pain perception in children.

ELIGIBILITY:
Inclusion Criteria:

* In need of treatment of right and left primary molar teeth of maxilla,
* Does not have any systemic disorder,
* High level of communication that can provide logical answers to the questions we ask
* With parental consent,
* Volunteers who want to participate in the research
* 6-12 years old patients who are compatible with routine dental treatments in the pediatric clinic

Exclusion Criteria:

* No need for treatment of right and left primary molar teeth of maxilla,
* Has a systemic condition
* Low level of communication that cannot provide reasonable answers to the questions we ask
* Without parental consent
* Do not want to participate voluntarily in the research
* Do not attend a check-in
* Patients not in the 6-12 age group

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale (PRS) | 3 months
  The PRS measures the unpleasantness or affective dimension of a child's pain experience and is used in children aged 3-17 years old. The PRS consists of a set of cartoon faces with varying facial expressions ranging from a smile/laughter to tears, and each child is asked to select the facial expression that best represents his/her experience of discomfort. Each face has a numerical value ranging from 0 (smiling face, "no hurt") to 5 (crying/screaming face, "hurts worst").
Face, Legg, Cry, Consolability Scale (FLACC) | 3 months
  The scale comprised the following parameters: (1) Face, (2) Legs, (3) Activity, (4) Cry, and (5) Consolability. Each of the five categories is scored from 0-2, which results in a minimum total score of 0 and maximumof 10. According to this scale: 0=Relaxed and comfortable (no pain); 1-3=Mild discomfort; 4-6=Moderate pain; and 7-10=Severe discomfort or pain [Willis et al., 2003]. Behavioural parameters were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No